CLINICAL TRIAL: NCT07060066
Title: Bilateral Prefrontal and Insular TMS for Depression in Schizophrenia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Xiaoming Du, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-MS-25-0607
Record Dates: First submitted 2025-07-01; First posted 2025-07-11 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia and Related Disorders
Keywords: transcranial magnetic stimulation; schizophrenia; depression
MeSH Terms: conditions — Schizophrenia; Depression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active rTMS stimulation (Active Comparator): Participants will receive active H-coil delivered rTMS in each treatment visit for up to 20 treatment visits for about 4 weeks. In each visit, there are three rTMS sessions with inter-rTMS-session interval of about 30 minutes.
  Interventions: Device: Active rTMS stimulation
- Sham rTMS stimulation (Sham Comparator): Participants will receive sham H-coil delivered rTMS in each treatment visit for up to 20 treatment visits for about 4 weeks. In each visit, there are three rTMS sessions with inter-rTMS-session interval of about 30 minutes.
  Interventions: Device: Sham rTMS stimulation

INTERVENTIONS:
Device: Active rTMS stimulation — Active H-coil delivered rTMS sessions will be given three times per treatment visit for up to 20 visits for about 4 weeks. There are about 30 minutes breaks between adjacent TMS sessions. Each TMS session takes about 3 to 4 minutes to complete.
  Arms: Active rTMS stimulation
Device: Sham rTMS stimulation — Sham H-coil delivered rTMS sessions will be given three times per treatment visit for up to 20 visits for about 4 weeks. There are about 30 minutes breaks between adjacent TMS sessions. Each TMS session takes about 3 to 4 minutes to complete.
  Arms: Sham rTMS stimulation

SUMMARY:
The purpose of this study is to provide an effective repetitive transcranial magnetic stimulation (rTMS) treatment for depressive symptoms in patients with schizophrenia. Schizophrenia patients with depressive symptoms will be exposed to rTMS to improve their symptoms.

DETAILED DESCRIPTION:
Schizophrenia spectrum disorder (SSD) and major depressive disorder (MDD) are often debilitating conditions, and thus not surprising that many SSD patients with comorbid depression have even poorer quality of life, higher suicide risk, worse clinical outcome, and higher rates of re-hospitalization than just having SSD alone. SSD patients with depression (DIS) suffered the unfortunate 'double whammy' by two of the most severe symptom categories in mental health.

Transcranial magnetic stimulation (TMS) is a non-invasive means for safely introducing the brain with electrical neural activity through magnetic stimulation on specific locations. Thousands of patients with depression and other psychiatric conditions have benefited from TMS through FDA-approved TMS devices. However, no TMS trial report has directly targeted DIS. The H4 coil is FDA-cleared to be marketed as deep TMS for short-term smoking cessation. This H4 coil targets bilateral insula and prefrontal cortices, which may underlie the depressive symptoms in SSD.

The patients with schizophrenia who also have depressive symptoms will receive rTMS via the H4 coil. The efficacy of using H4 rTMS for treating depressive symptoms in schizophrenia patients will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male and female ages between ages 18-60 years.
* Ability to give written informed consent (age 18 or above).
* Diagnosed with schizophrenia-spectrum disorder and Evaluation to Sign Consent (ESC) above 10.
* Score of Calgary depression scale for schizophrenia (CDSS) ≥ 3.

Exclusion Criteria:

* Inability to sign informed consent.
* Any major medical illnesses that may affect normal brain functioning. Examples of these conditions include, but are not limited to: stroke, repeated seizure, history of significant head trauma with cognitive sequela, CNS infection or tumor, other significant brain neurological conditions.
* Significant alcohol or other drug use other than nicotine or marijuana dependence.
* Inability to refrain from using alcohol and/or marijuana 24 hours or more prior to experiments.
* Pregnancy, as classified by a woman of child-bearing potential who is not using a contraceptive and has missed a menstrual period; or by self-report; or by positive urine pregnancy test.
* For MRI, inability to participate in the MRI scanning due to metallic devices or objects (cardiac pacemaker or neurostimulator, some artificial joints, metal pins, surgical clips or other implanted metal parts) or declining to get in the scanner.
* Failed TMS safety questionnaire.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2030-06-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Brain connectivity as indicated by resting-state functional connectivity (rsFC) values as assessed by functional MRI (fMRI) | baseline, visit 11 (about 2 week after baseline), visit 21 (about 4 weeks after baseline)
  rsFC values will be reported as a Z-score with a range of -1 to 1, with greater absolute values indicating stronger brain connectivity.

SECONDARY OUTCOMES:
Electrophysiological response as indicated by mismatch negativity as assessed by electroencephalography (EEG) | baseline, visit 11 (about 2 week after baseline), visit 21 (about 4 weeks after baseline)
  Mismatch negativity values will be reported in microvolts (uV). Mismatch negativity is measured by subtracting the averaged response to a set of standard stimuli from the average response to deviant stimuli, and taking the amplitude of this difference in a given timepoint.
Electrophysiological response as indicated by steady-state auditory evoked responses from electroencephalography recording (EEG) | baseline, visit 11 (about 2 week after baseline), visit 21 (about 4 weeks after baseline)
  Steady-state auditory evoked responses will be reported. The responses are measured by calculating the ratio of the power at target frequency over power at the surrounding background frequencies. The ration will be obtained in a given timepoint.
Depression as assessed by the Calgary Depression Scale | baseline, visit 11 (about 2 week after baseline), visit 21(about 4 weeks after baseline)
  Total score of the Calgary Depression Scale will be reported and ranges from 0 to 27, with a higher score indicating greater depression.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoming Du, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No